CLINICAL TRIAL: NCT06568484
Title: Bedaquiline Roll-out Evidence in Contacts and People Living With HIV to Prevent TB (BREACH-TB)
Brief Title: Bedaquiline Roll-out Evidence in Contacts and People Living With HIV to Prevent TB
Acronym: BREACH-TB
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other); US Department of State (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00443418; 7200AA22CA00005 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis, Latent
Keywords: Bedaquiline
MeSH Terms: conditions — Latent Tuberculosis | interventions — bedaquiline; Isoniazid; rifapentine; Levofloxacin

STUDY DESIGN:
Intervention Model Description: A seamless, staged, Phase II/III, open-label, multicenter, noninferiority trial to compare the efficacy and safety of 4 weeks of oral bedaquiline (1BDQ) versus a standard regimen for preventing confirmed or probable tuberculosis disease (TBD) during 72 weeks of follow-up among people living with HIV (PLHIV) and high-risk Close Contacts (CC) of Index Patients with Drug-Susceptible (DS) or Rifampin-Resistant (RR) TB. CCs that are also household contacts will be cluster-randomized by household.
  The study will be divided into two stages, with a seamless transition between stages, meaning enrollment into Stage 2 will start while Stage 1 outcomes analyses are ongoing. All recruited patients will be followed up to 72 weeks post randomization.
Who Masked: Outcomes Assessor
Masking Description: An independent Endpoint Review Committee (ERC), masked to study arm, will adjudicate the incident TB endpoints (both primary and secondary) and, if there are any deaths, determine the cause of death as TB-related or not TB-related.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bedaquiline (Experimental): 4 weeks of daily bedaquiline
  Interventions: Drug: Bedaquiline
- 3HP (Active Comparator): 3 months of weekly isoniazid (H) and rifapentine (P)
  Interventions: Combination Product: Isoniazid, rifapentine
- Levofloxacin (Active Comparator): 6 months of daily levofloxacin
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Bedaquiline — CCs (Close Contacts) of DS-TB Index Patients and PLHIV at high risk of developing TBD
  1. Children 0 to <5 years old who are HIV negative, regardless of latent tuberculosis infection (LTBI) result by TST (tuberculin skin test) or IGRA (interferon-gamma release assay)
  2. Adults, pregnant people, adolescents, and children ≥5 years old who are HIV negative and LTBI positive (by IGRA)
  3. Adults and adolescents ≥15 years of age who are living with HIV regardless of LTBI status, regardless of whether the participant is a CC
  CCs of RR-TB Index Patients at high risk of developing TBD
  1. Children 0 to <5 years old, regardless of HIV status or LTBI result (by TST or IGRA)
  2. Adults, adolescents, and children ≥5 years old who are HIV negative and LTBI positive (by IGRA)
  3. Adults, pregnant people, adolescents, and children ≥5 years old who are living with HIV regardless of LTBI status
  Bedaquiline based on weight and/or age at Enrollment daily for four weeks (28 doses)
  Other Names: Sirturo
  Arms: Bedaquiline
Combination Product: Isoniazid, rifapentine — CCs of DS-TB Index Patients and PLHIV at high risk of developing TBD
  1. Children 0 to <5 years old who are HIV status negative, regardless of latent tuberculosis infection (LTBI) result (WHO-recommended skin test or interferon-gamma release assay [IGRA])
  2. Adults, adolescents, and children ≥5 years old who are HIV status negative and LTBI positive (by IGRA)
  3. Adults and adolescents ≥15 years of age who are living with HIV regardless of LTBI status, regardless of whether they are a CC
  3HP: 3 months of weekly isoniazid (H) and rifapentine (P) (12 doses)
  Other Names: 3HP
  Arms: 3HP
Drug: Levofloxacin — CCs of RR-TB Index Patients at high risk of developing TBD
  1. Children 0 to <5 years old, regardless of HIV status or LTBI result (by TST or IGRA)
  2. Adults, adolescents, and children ≥5 years old who are HIV status negative and LTBI positive (by IGRA)
  3. Adults, pregnant people, adolescents, and children ≥5 years old who are living with HIV regardless of LTBI status
  Levofloxacin (LFX) based on weight at Enrollment daily for 6 months (182 doses)
  Other Names: Levaquin
  Arms: Levofloxacin

SUMMARY:
A seamless, staged Phase II/III, open-label, multicenter, non-inferiority trial, to compare the efficacy and safety of 4 weeks of bedaquiline (BDQ) versus a a standard regimen for preventing regimen for preventing confirmed or probable tuberculosis disease (TBD) during 72 weeks of follow-up among people living with HIV (PLHIV) and high-risk Close Contacts (CC) of adults with Drug Susceptible (DS) or Rifampin Resistant (RR) TB.

DETAILED DESCRIPTION:
Treating adult, adolescent, child, and pregnant close contacts (CCs) of drug-sensitive tuberculosis (DS-TB) who are high-risk for developing tuberculosis disease (TBD) as well as adult and adolescent people living with HIV (PLHIV) in high-tuberculosis burden regions with bedaquiline (BDQ) will be noninferior in reducing the risk of developing TBD compared with a WHO-recommended rifamycin-containing short-course regimen for TB preventive therapy (TPT).

Treating adult, adolescent, child, and pregnant CCs of rifampin-resistant tuberculosis (RR-TB) who are high-risk for developing TBD with BDQ will be noninferior in reducing the risk of developing TBD compared with levofloxacin.

ELIGIBILITY:
INCLUSION CRITERIA

For Index Patient

• Any age

* A diagnosis of bacteriologically proven pulmonary TB
* Initiated on treatment for pulmonary TB within the past 90 days
* Have at least one close contact that is likely to be eligible for the study

For PLHIV Indication

Individuals must meet all of the following inclusion criteria to participate in this study:

* On a dolutegravir-based or other approved integrase inhibitor antiretroviral therapy (ART) regimen that does not interact with bedaquiline or rifapentine.

  * If on a protease inhibitor-based ART regimen, a participant can be enrolled following a 5-day washout with switch to a dolutegravir-based regimen prior to enrollment. A 14-day washout is required for efavirenz-based ART regimen with switch to a dolutegravir-based regimen prior to enrollment
  * If a participant is not currently on ART or is ART-naïve, the participant must have started a dolutegravir-based ART regimen prior to Enrollment.
* PLHIV who meet criteria for a TBD close contact should be enrolled under the close contact indication

For Close Contact Indication (DS- or RR-TB Index Patient)

* Definition of Close Contact (either/or):

  o Lives or lived in the same dwelling unit or plot of land and shares or has shared the same housekeeping arrangements as the Index Patient for one or more nights ≤ 90 days prior to the Index Patient starting TB treatment

  o Has shared more than four hours of indoor airspace with the Index Patient during any one-week period ≤ 90 days prior to the Index Patient starting TB treatment. This may include indoor airspace within or outside the home.
* Close contacts must be in one of the following high-risk groups:

  * All children 0 to <5 years old at the time of Enrollment, regardless of LTBI or HIV status
  * Adults, adolescents, and children ≥5 years of age who are TBI test positive (either skin test positive* or IGRA-positive) and whose HIV status is negative, indeterminate, or unknown.
  * Adults, adolescents, and children ≥5 years of age who have a documented HIV infection regardless of TBI test status.

Universal Enrollment Inclusion Criteria for PLHIV and Close Contacts of DS- or RR-TB Index Patient

A. Ability and willingness of participant (and/or parent/guardian) to provide informed consent (and assent, as applicable)

B. Documentation of HIV Status

For participants >=18 months of age known to be PLHIV:

* Certified copy of HIV clinic card or
* Certified copy of HIV testing that includes date, assay used and result

For participants <18 months of age who have never tested, or previous HIV test result was indeterminate, unknown, or negative more than three months prior to screening and/or result is not available:

• HIV-1 testing should be performed per Section 5.4.5 (HIV-1 Testing) during the study screen period.

For participants <18 months known to be CLHIV:

• Certified copies of HIV DNA and/or RNA testing that includes date, assay used, and result

For participants <18 months who have never tested, or previous HIV test result was indeterminate, unknown, or negative more than three months prior to screening and/or result is not available:

• HIV-1 testing should be performed per Section 5.4.5 (HIV-1 Testing) during the study screen period

C. Documentation of ART

* All PLHIV (for PLHIV indication and CC that are PLHIV) must be on a dolutegravir-based or other approved integrase inhibitor ART regimen that does not interact with bedaquiline or rifapentine.
* If on a protease inhibitor-based ART regimen, a participant can be enrolled following a 5-day washout with switch to a dolutegravir-based regimen prior to enrollment. A 14-day washout is required for efavirenz-based ART regimen with switch to a dolutegravir-based regimen prior to enrollment.
* If a participant is not currently on ART or is ART-naïve, they must have started a dolutegravir-based ART regimen prior to Enrollment.

D. Chest radiograph without evidence of active TBD, performed within 30 days prior to Enrollment

E. The following laboratory values obtained within 30 days prior to Enrollment.

* Alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal
* Total bilirubin ≤ 2.5 times the upper limit of normal
* Alkaline phosphatase ≤ 3 times the upper limit of normal
* Creatinine clearance ≥ 29 ml/min
* Serum potassium at or above the lower limit of normal
* Serum magnesium at or above the lower limit of normal
* Serum calcium at or above the lower limit of normal
* Platelet count of ≥ 50,000 /mm3
* Absolute neutrophil count (ANC) ≥ 1,000/mm3

F. Pregnancy test (for study candidates of childbearing potential*)

• Negative serum or urine pregnancy test within 7 days prior to enrollment.

*NOTE: Participants of childbearing potential are defined as females who have reached menarche or who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) or have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).

EXCLUSION CRITERIA

Exclusion Criteria for Index Patient A. Unwilling or unable to provide informed consent B. No close contacts likely to be eligible for the study C. Study staff unable to obtain status of TB drug susceptibility or resistance D. Known bedaquiline resistance of M. tb isolate E. Known fluoroquinolone resistance of M. tb isolate (for Index Patients with RR-TB)

Exclusion Criteria for PLHIV and Close Contacts of DS- or RR-TB Index Patient

A. Unwilling or unable to provide informed consent

B. Weight ≤ 3 kg

C. A current diagnosis of confirmed or probable or possible pulmonary or extrapulmonary TB at time of enrollment or confirmed or unconfirmed TB for children.

D. Previously completed treatment for TBD.

E. Prior completion of TPT (including but not limited to 6 or 9H, 1HP, 3HP, 4R, 3HR, 6Lfx) *

*NOTE: Completion of TBD treatment or TPT based on the opinion of the site investigator that a sufficient course of TPT was taken to constitute treatment completion

F. Current enrollment into another therapeutic clinical trial (See Section 5.8).

G. Any of the following medical conditions:

* Severe renal impairment (DAIDS Grade 4) or end-stage renal disease requiring hemodialysis or peritoneal dialysis
* Severe hepatic impairment (Child-Pugh C)
* Evidence of acute hepatitis, such as abdominal pain, jaundice, dark urine, and/or light stools within 90 days prior to enrollment
* Severe cardiac arrythmia requiring medication
* Peripheral neuropathy ≥ Grade 2 (DAIDS)
* Diagnosis of porphyria at any time prior to study enrollment
* Corrected QTcF (Fridericia's formula) of >460 msec
* Unable to take oral medication
* Active drug or alcohol use or dependence that, in the site investigator's opinion, would interfere with adherence to study treatment.
* Serious illness requiring systemic treatment including parenteral therapy (e.g., antibiotics) and/or hospitalization within 30 days prior to Enrollment
* Prior exposure to bedaquiline or clofazimine
* Receipt of more than 7 cumulative days of isoniazid, a rifamycin, or a fluoroquinolone in the 90 days prior to enrollment
* Known bedaquiline resistance in Index Patient
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
* Currently taking another medication that is prohibited with study medicines which cannot be stopped (with or without replacement) or requires a washout period longer than 14 days (See Appendix 7)
* Known pregnancy or breastfeeding

Specific Exclusion Criteria for Close Contacts of RR-TB Index Patient

* Known fluoroquinolone resistance in Index Patient
* Severe tendinopathy related to fluoroquinolones

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2530 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety DS-TB CCs and PLHIV (Stage 1): Proportion of participants who permanently discontinue the randomized study drug due to a treatment-related adverse event by 18 weeks | 18 weeks
  Estimate of the safety of 1BDQ and 3HP among adult, adolescent, and child CCs of DS-TB Index Patients at high risk of developing TBD, as well as adult and adolescent PLHIV in high TB-burden settings
Safety for RR-TB CCs (Stage 1): Proportion of participants who permanently discontinue the randomized study drug due to a treatment-related adverse event by 36 weeks | 36 weeks
  Estimate of the safety of 1BDQ and 6 months of levofloxacin (6L) among adult, adolescent, and child CCs of RR-TB Index Patients at high risk of developing TBD
Treatment Completion - PLHIV & CCs of DS-TB (Stage 1): Proportion of participants completing assigned treatment within window prescribed in protocol | 18 weeks
  Estimate on-time treatment completion of 1BDQ & 3HP in adult, adolescent, & child CCs of DS-TB Index Patients at high risk of developing TBD, & adult and adolescent PLHIV in high TB-burden countries
Treatment Completion - CCs of RR-TB (Stage 1): Proportion of participants completing assigned treatment within window prescribed in protocol | 36 weeks
  Estimate on-time treatment completion of 1BDQ and 6 months of levofloxacin (6L) among adult, adolescent, and child CCs of RR-TB Index Patients at high risk of developing TBD
Primary Efficacy Endpoint (Stage 2): Number of enrolled participants (PLHIV, contacts of DS-TB or RR-TB) diagnosed with bacteriologically confirmed or probable / (if adult), and confirmed or unconfirmed (if child) TB disease | Up to 72 weeks post-treatment initiation
  Number (per person-years) of participants diagnosed with confirmed or probable (if adult) and unconfirmed or confirmed (if child) TB disease, compared between the comparator arm and investigational (BDQ) arm and expressed as the averted events ratio (AER)
Primary Safety Endpoint (Stage 2): Cumulative number of enrolled participants (PLHIV, contacts of DS-TB or RR-TB) who permanently discontinue the assigned study regimen due to an adverse drug reaction | Varies by treatment regimen (1 month, 3 months, or 6 months)
  Proportion of individuals who permanently discontinue assigned study regimen due to a treatment-related adverse event, compared between the comparator arm and investigational (BDQ) arm.

SECONDARY OUTCOMES:
Stage 1: Proportion of participants who permanently discontinue the randomized study drug due to a treatment-related adverse event by 18 weeks | 18 weeks
  To compare the safety of 1BDQ to 3HP among adult, adolescent, and child CCs of DS-TB Index Patients at high risk of developing TBD as well as adult and adolescent PLHIV in high TB-burden settings
Stage 1: Proportion of participants who permanently discontinue the randomized study drug due to a treatment-related adverse event by 36 weeks | 36 weeks
  To compare the safety of 1BDQ to 6 months of levofloxacin (6L) among adult, adolescent, and child CCs of RR-TB Index Patients at high risk of developing TBD
Stage 1: Proportion of participants completing assigned treatment within window prescribed in protocol | Dependent on treatment assignment (1 month, 3 months, or 6 months)
  To compare on-time treatment completion of 1BDQ to 6 months of levofloxacin (6L) among adult, adolescent, and child CCs of RR-TB Index Patients at high risk of developing TBD
Stage 1: Proportion of individuals who experience a grade 3 or higher AE, compared between the comparator arm and investigational (1BDQ) arm at 18 weeks | 18 weeks
  To compare the safety of 1BDQ to 3HP among adult, adolescent, and child CCs of DS-TB Index Patients at high risk of developing TBD, as well as adult and adolescent PLHIV in high TB-burden settings
Stage 1: Proportion of participants completing assigned treatment within window prescribed in protocol | Dependent upon treatment assignment (1 month, 3 months, or 6 months)
  To compare on-time treatment completion of 1BDQ to 3HP among adult, adolescent, and child CCs of DS-TB Index Patients at high risk of developing TBD as well as adult and adolescent PLHIV in high TB-burden settings
Stage 1: Proportion of individuals who experience a grade 3 or higher AE, compared between the comparator arm and investigational (1BDQ) arm at 36 weeks | 36 weeks
  To compare the safety of 1BDQ to 6 months of levofloxacin (6L) among adult, adolescent, and child CCs of RR-TB Index Patients at high risk of developing TBD
Stage 1: Proportion of participants who experience a TBD event at up to 72 weeks of follow-up, by study arm | Up to 72 weeks
  To estimate the number of incident TBD events in each study arm, at up to 72 weeks of follow-up
Secondary Efficacy Endpoint (Stage 2): # of enrolled participants (PLHIV, contacts of DS-TB, RR-TB) who reach a composite outcome of bacteriologically confirmed, probable, or possible (if adult) and confirmed or unconfirmed (if child) TBD or death | 72 weeks post-treatment initiation
  Number, per person-years, of participants diagnosed with bacteriologically confirmed, probable, or possible (if adult) and confirmed or unconfirmed (if child) TB disease or death from any cause (except for violent or accidental death), compared between the comparator arm and investigational (BDQ) arm and expressed as the AER.
Secondary Safety Endpoint (Stage 2): Cumulative number of enrolled participants (PLHIV, contacts of DS-TB or RR-TB) who experience a grade 3 or higher AE | Varies by treatment regimen duration (1 month, 3 months, or 6 months)
  Proportion of individuals who experience a grade 3 or higher AE, compared between the comparator arm and investigational (BDQ) arm
Secondary Endpoint of Treatment Completion (Stage 2): Proportion of participants who have taken at least 90% of the doses within the specified timeframe of the assigned regimen | Varies by treatment regimen duration (1 month, 3 months, or 6 months)
  The absolute difference in proportions of the number of participants who have taken at least 90% of their doses within the specified timeframe of their assigned regimen, and the corresponding 95% confidence interval
Stage 1: Proportion of participants who experience a composite outcome at up to 72 weeks of follow-up, by study arm | Up to 72 weeks
  To estimate the number of composite outcomes of confirmed, probable or possible (if adult), or confirmed or unconfirmed (if child) TBD & all-cause mortality due to any cause, except violent or accidental death in each study arm, up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Nuermberger, MD, Study Chair — Johns Hopkins School of Medicine
Locations (6):
- Peru (2):
  - HNSEB (Hospital Nacional Sergio E. Bernales), Lima
  - SES Policlinico, Lima
- Kilimanjaro Clinical Research Institute, Moshi, Tanzania
- Uganda (3):
  - Joint Clinical Research Centre, Kampala
  - Makerere Lung Institute, Kampala
  - MU-JHU Care Ltd., Kampala

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that can be legally released.
Supporting Information: Study Protocol, SAP, ICF